CLINICAL TRIAL: NCT05769322
Title: Remote Electrical Neuromodulation (REN) Wearable Device for Adolescents with Migraine: Real World Study of High-Frequency Users Suggest Preventive Effects
Brief Title: Real World Data Analysis: Impact of High-Frequency REN Treatments As Migraine Preventive Therapy in Adolescence
Status: Completed | Type: Observational
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Other Study IDs: RWE005
Record Dates: First submitted 2023-03-02; First posted 2023-03-15 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2023-02

CONDITIONS: Migraine
Keywords: Migraine prevention; headache; Nerivio; REN
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Nerivio — Remote electrical neuromodulation (REN) device for the acute treatment of migraines. The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application.

SUMMARY:
This is a post-marketing study investigating the safety and efficacy of the REN device (Nerivio by Theranica, ISRAEL) in adolescents with migraine. The data analysis will test the ability of Frequent use of REN for the acute treatment of migraine to reduce the number of monthly migraine days in subsequent months, suggesting potential preventive benefits.

DETAILED DESCRIPTION:
The REN device (Nerivio by Theranica, ISRAEL) is a neuromodulation device approved by the FDA for acute and/or preventive treatment of migraine in patients of 12 years old and above. It is a wearable device applied to the upper arm. It stimulates C and Aδ noxious fibers using a modulated, symmetrical, biphasic, square pulse with a pulse width of 400 μs, modulated frequency of 100-120 Hz, and up to 40 mA output current which the patient can adjust. The REN device is operated by a designated app that is downloaded to the user's phone prior first use of the Nerivio device.

As part of the sign-up process to the Nerivio app, all patients accept the terms of use which specify that providing personal information is done by their own free will and that their de-identified data may be used for research purposes. Users are not obligated to provide personal information and could treat without providing any feedback. The app includes a secured, personal migraine diary, which enables patients to record and track their migraines and other headaches. At the beginning of each treatment, and again 2 hours after the start of treatment, patients are prompted to record their symptoms, including pain level (none, mild, moderate, severe), functional disability (No limitation, Some limitation, Moderate limitation, Severe limitation), and an indication of which medications, if any, were taken within that 2-hour time window.

This post-marketing RWE study investigates the potential of high usage of Nerivio for the acute treatment of migraine on migraine prevention, using the following outcomes:

1. - reduction in mean monthly migraine treatment days (MMTD),
2. - acute treatment efficacy measured 2 h post-treatment
3. - improve in functional disability
4. - Device safety

Together, these objectives may provide a comprehensive evaluation of the impact of the high usage of Nerivio for acute treatment as a migraine preventive tool in the migraine adolescent population.

ELIGIBILITY:
Inclusion Criteria:

* patient age is 12 Years to 18 Years
* Patient is using the Nerivio device for acute treatment of migraine
* Patient treated at least 10 treatments in his first month of using Nerivio and at least 3 treatments in each of the two consecutive months (months 2 and 3

Exclusion Criteria:

* Treatments shorter than 30 minutes

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescence (age 12-18) who suffers from migraine and are using the Nerivio device for acute treatment of migraine.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Reduction in Mean Monthly Migraine Treatment Days | 3 months
  Mean number of migraine treatment days per month during 3 consecutive months, comparing each month to the first month.
  A migraine treatment day is defined as a day in which a patient treated their migraine with REN.

SECONDARY OUTCOMES:
Consistent Headache Relief at 2 Hours Post-treatment | 2 hours
  The proportion of subjects reporting headache relief at 2 hours post-treatment in at least 50% of all their treatments.
  headache relief is defined as an improvement from severe or moderate pain to mild or no pain. Pain level is reported using a 4-point Likert scale (0 - No pain, 1 - Mild pain, 2 - Moderate pain,3- Severe pain)
Consistent Freedom From Headache at 2 Hours Post-treatment | 2 hours
  The proportion of subjects reporting freedom from headache at 2 hours post-treatment in at least 50% of all their treatments. Pain freedom is defined as the disappearance of headache from severe, moderate, or mild headache at treatment initiation to no headache 2 hours later.
  Pain level is reported using a 4-point Likert scale (0 - No pain, 1 - Mild pain, 2 - Moderate pain,3- Severe pain).
Consistent Functional Disability Relief at 2 Hours Post-treatment | 2 hours
  The proportion of subjects who reported having Functional Disability at the beginning of the treatment and reported improvement of at least one level of Functional Disability at 2 hours post-treatment in at least 50% of all their treatments.
  Functional Disability level is reported using a 4-point Likert scale (0 - No limitation, 1 - Some limitation, 2 - Moderate limitation, 3 - Severe limitation).
Consistent Functional Disability disappearance at 2 Hours Post-treatment | 2 hours
  The proportion of subjects who reported having Functional Disability at the beginning of the treatment and reported no Functional Disability at 2 hours post-treatment in at least 50% of all their treatments.
  Functional Disability level is reported using a 4-point Likert scale (0 - No limitation, 1 - Some limitation, 2 - Moderate limitation, 3 - Severe limitation).
Device Related Adverse Events | 3 months
  Incidence of device-related adverse events reported by subjects

CONTACTS AND LOCATIONS:
Overall Officials: Alit Stark Inbar, PhD, Principal Investigator — Theranica Bio-Electronics Ltd
Locations (1):
- Theranica USA Inc, Bridgewater, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No